CLINICAL TRIAL: NCT06740656
Title: Neuromuscular Complications of MEK Inhibitors: a French Case Series and a Systematic Review of the Literature
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pauline DUCATEL, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2024PI240
Record Dates: First submitted 2024-12-08; First posted 2024-12-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Myositis; Myasthaenia Gravis; Neuropathy; Guillain Barré Syndrome; Parsonage Turner Syndrome
MeSH Terms: conditions — Myositis; Guillain-Barre Syndrome; Brachial Plexus Neuritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Interventions — no intervention

SUMMARY:
MEK inhibitors (trametinib, cobimetinib, selumetinib or binimetinib) have been used since 2016 to treat metastatic melanoma, by targeting the MAPK pathway Neuromuscular complications (neuropathy, myasthenia or myositis) have been reported in patients treated with MEK inhibitors.

With the growing use of these new oncology therapies, neurologists, oncologists and other clinicians are likely to be increasingly confronted with MEK inhibitor-induced neuropathy, myasthenia or myositis.

Yet, so far, these complications have only been documented in a few single case reports.

Our aim was to characterize the neuromuscular complications associated with MEK inhibitors used either alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuromuscular complications of MEK inhibitors used alone or in combination
* Age > 18 years

Exclusion Criteria:

* Refusal of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuromuscular complications treated with MEK inhibitors at a Neuromuscular Reference Center in France
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Type of neuromuscular complications | up to 8 years

SECONDARY OUTCOMES:
Time to onset after introduction of MEK inhibitors | up to 8 years
Severity of neuromuscular complications | up to 8 years
Progression with or without treatment | up to 8 years
Reintroduction of MEK inhibitors | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Ducatel, Doctor, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France